CLINICAL TRIAL: NCT04087889
Title: Individual Patient Expanded Access IND of Hope Biosciences Allogeneic First Blood Relative Adipose-derived Mesenchymal Stem Cells (HB-adMSCs) for Pancreatic Cancer
Brief Title: Individual Patient Expanded Access IND of Hope Biosciences First Blood Relative Allogeneic Adipose-derived Mesenchymal Stem Cells (HB-adMSCs) for Pancreatic Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences LLC (Industry)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Other Study IDs: HBPC01
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: Cancer; Pancreas; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Adenocarcinoma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — Culture-expanded, adipose-derived mesenchymal stem cells donated by first blood relative

SUMMARY:
The drug for this submission is Hope Biosciences' allogeneic, first blood relative, adipose-derived culture-expanded mesenchymal stem cells (HB-adMSCs) for the treatment of a single patient with Pancreatic Cancer (PC). PC is an extremely infiltrative neoplasm that usually presents with vascular and perineural invasion in surgically resected tumors. Metastases to lymph nodes, liver and distant sites are all very common. Its incidence has markedly increased over the past several decades and ranks as the fourth leading cause of cancer death in the United States. Despite the high mortality rate associated with pancreatic cancer, its etiology is poorly understood. PC patients experience physiological symptoms such as anemia, ascites, severe fatigue, pain, cachexia, weakness, insomnia, confusion, and memory loss. The aggressive nature of PC leads to rapid deterioration of patients' quality of life and diminished ability to participate in treatment.

DETAILED DESCRIPTION:
Once the eligibility is confirmed, approximately 1-3 weeks after the screening/baseline visit, the subject will return for the first infusion. Subsequent treatments will occur weekly for the first 8 infusions, followed by 4 infusion that occur 2 weeks apart. The total number of infusions will be 12.

On each of these visits, the subject will receive one allogeneic HB-adMSC infusion of 200 million (2 x 10^8 cells) total cells suspended in 250 mL normal saline for IV infusion. Every infusion visit will include the following procedures:

1. Review of medical history,
2. Complete Physical exam (Week 1, 4, 10, 20, and 52),
3. Vital signs (Heart Rate, BP, Respirations, Temp., SpO2),
4. Weight measurement
5. A verification of patient consent will be verbally performed
6. *When applicable (Week 4, 7, 10, 14, 20 and 52): A urine and blood sample for clinical labs including:

   * CBC with diff.,
   * CMP,
   * Coagulation Panel,
   * TNF-a
   * IL-6
   * CA 19-9
   * LDH
7. The HB-adMSC infusion will be given via IV.
8. The subject will then be monitored for a minimum of 2hr after infusion.
9. 24-hour telephone assessment for adverse events
10. Video Documentation

Vital signs will be continuously monitored during the infusion and recorded at 15 minutes intervals during the first hour. Vital signs will be recorded at the end of the infusion and every 30 minutes x 2 hours or more frequently if clinically indicated. The subject will be contacted by telephone 24hr. after the infusion visit to determine if any adverse events have occurred.

*Please note that blood and urine sample during the intervention period will only be required for the visits corresponding to weeks 4, 7, 10, 14, 20 and 52. During these visits, these samples will always be taken before the infusion is started. Refer to Table 1. Schedule of assessments for more details.

Follow-up Visits week 4,7, 10, 14, 20, and 52

The subject will undergo the following procedures at each follow-up visit without infusion:

1. Review and update medical history,
2. Update concomitant medications list
3. Weight
4. Vital signs (Heart Rate, BP, Respirations, Temp., SpO2),
5. Complete physical exam (Week 1, 4, 10, 20, and 52)
6. A urine and blood sample for clinical labs including:

   * CBC with diff.,
   * CMP,
   * Coagulation Panel,
   * TNF-a
   * IL-6
   * CA 19-9
   * LDH
7. Adverse event monitoring.

In addition, visits 13 and 14 (week 20 and 52) will include CT Scans of the chest, abdomen and pelvis. This procedure could be done up to 7 days before or after the actual visit day, depending on availability and schedule of the imaging center. If a CT Scan has been done as standard of care within 30 days of these visits, it would meet the requirement for this assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Pancreatic Cancer
2. Hemodynamically stable

Exclusion Criteria:

1. Immunosuppression as defined by WBC < 3, 000 cells/ml at baseline screening.
2. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSC administration.
3. Any abnormal, inexplicable laboratory result with no obvious cause defined.
4. Participation in other interventional research studies. Unwillingness to return for follow-up visits

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Biosciences, Sugar Land, Texas, United States